CLINICAL TRIAL: NCT01621178
Title: A Randomized, Open-Label, Parallel-Arm Study Comparing the Effect of Once-weekly Dulaglutide With Insulin Glargine on Glycemic Control in Patients With Type 2 Diabetes and Moderate or Severe Chronic Kidney Disease
Brief Title: A Study Comparing Dulaglutide With Insulin Glargine on Glycemic Control in Participants With Type 2 Diabetes (T2D) and Moderate or Severe Chronic Kidney Disease (CKD)
Acronym: AWARD-7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13798; H9X-MC-GBDX (Other: Eli Lilly and Company); 2012-000829-44 (EudraCT Number)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — dulaglutide; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Masking Description: Dulaglutide dose was blinded to participant, care provider, investigator and outcomes assessor.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin glargine (Active Comparator): Insulin glargine was administered subcutaneously (SC) at bedtime per a modified forced-titration treat-to-target algorithm. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
  Interventions: Drug: Insulin glargine; Drug: Insulin lispro
- 0.75 mg Dulaglutide (Experimental): 0.75 milligram (mg) of dulaglutide was administered once weekly as a SC injection. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
  Interventions: Drug: Dulaglutide; Drug: Insulin lispro
- 1.5 mg Dulaglutide (Experimental): 1.5 mg of dulaglutide was administered once weekly as a SC injection. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
  Interventions: Drug: Dulaglutide; Drug: Insulin lispro

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: 0.75 mg Dulaglutide; 1.5 mg Dulaglutide
Drug: Insulin glargine — Administered SC
  Arms: Insulin glargine
Drug: Insulin lispro — Administered SC

SUMMARY:
The purpose of this study is to determine the glycemic efficacy and safety of dulaglutide compared to insulin glargine in the treatment of participants with type 2 diabetes and moderate or severe chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women aged ≥18 years
* Hemoglobin A1c (HbA1c) ≥7.5% and ≤10.5%
* Type 2 diabetes on insulin or insulin + oral antihyperglycemic medication
* Participants with presumed diabetic kidney disease with or without hypertensive nephrosclerosis diagnosed with moderate or severe CKD with estimated glomerular filtration rate (eGFR) of ≥15 to <60 milliliters per minute (mL/min)/1.73 meter squared (m^2)
* Able and willing to perform multiple daily injections
* Body mass index (BMI) between 23 and 45 kilogram/square meter (kg/m^2)

Exclusion Criteria:

* Stage 5 CKD as defined by eGFR <15 mL/min/1.73 m^2 OR having required dialysis
* Rapidly progressing renal dysfunction likely to require renal replacement
* History of a transplanted organ
* Type 1 diabetes mellitus
* At screening a systolic blood pressure of ≥150 mmHg or a diastolic blood pressure of ≥90 mmHg with or without antihypertensive medication
* An episode of ketoacidosis or hyperosmolar state/coma in the past 6 months or a history of severe hypoglycemia in the past 3 months prior to the Screening Visit
* Cardiovascular conditions within 12 weeks prior to randomization: acute myocardial infarction, New York Heart Association (NYHA) class III or class IV heart failure, or cerebrovascular accident (stroke)
* Acute or chronic hepatitis
* Signs and symptoms of chronic or acute pancreatitis, or were in the past diagnosed with pancreatitis
* Serum calcitonin ≥35 picograms per milliliter (pg/mL) at Screening Visit
* Self or family history of medullary C-cell hyperplasia, focal hyperplasia, or carcinoma
* Known history of untreated proliferative retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2012-07; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (89):
- United States (47):
  - Extended Arm Physician, Inc., Montgomery, Alabama
  - North American Research Institute, Azusa, California
  - Renal Consultants Medical Group, Granada Hills, California
  - Marin Endocrine Associates, Greenbrae, California
  - Academic Medical Research Institute, Los Angeles, California
  - Sutter Gould Medical Foundation, Modesto, California
  - Infosphere, West Hills, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - The Center for Diabetes & Endocrine Care, Hollywood, Florida
  - East Coast Clinical Research, Jacksonville, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Avanced Medical and Pain Mangement Research Clinic (AMPM), Miami, Florida
  - Baptist Diabetes Association, Miami, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Discovery Medical Research Group, Ocala, Florida
  - Suncoast Clinical Research, Palm Harbor, Florida
  - University of Hawaii Clinical Research, Honolulu, Hawaii
  - Boise Kidney & Hypertension Institute, Caldwell, Idaho
  - Pacific Renal Research Institute, Meridian, Idaho
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Univ of Kansas Schl of Medicine , Wichita, Wichita, Kansas
  - Penobscot Bay Medical Center, Rockport, Maine
  - Nebraska Nephrology Research Institute, LLC, Lincoln, Nebraska
  - Endocrine Group, LLP, Albany, New York
  - Erie County Medical Center State University, Buffalo, New York
  - Institute for clinical studies, Rosedale, New York
  - Endocrine Associates of Long Island, PC, Smithtown, New York
  - Carolina Clinical Trials LLC, Concord, North Carolina
  - Physicians East, Greenville, North Carolina
  - Diabetes & Endocrinology Consultants PC, Morehead City, North Carolina
  - Boice Willis Clinic, PA, Rocky Mount, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Partners in Nephrology & Endocrinology, Pittsburgh, Pennsylvania
  - South Carolina Nephrology and Hypertension Center, Inc., Orangeburg, South Carolina
  - Carolina Diabetes & Kidney Ctr. Sumter Medical Specialist, Sumter, South Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Center For Clinical Research, Austin, Texas
  - Endocrine Associates of Dallas, Dallas, Texas
  - Office of Dr. Sergio Rovner, El Paso, Texas
  - Endocrine Associates, LLC, Houston, Texas
  - Juno Research, Houston, Texas
  - The Endocrine Center, Houston, Texas
  - San Antonio Kidney Disease Center Physicians Group, San Antonio, Texas
  - Providence Health & Services, Spokane, Washington
- Brazil (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belém
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Juiz de Fora
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Passo Fundo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Catarina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Hungary (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esztergom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaposvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kecskemét
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pécs
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sátoraljaújhely
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siófok
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Culiacán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zgierz
- Romania (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bacau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- South Africa (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johannesburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Ukraine (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Luhansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poltava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ternopil

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Tuttle KR, Lakshmanan MC, Rayner B, Busch RS, Zimmermann AG, Woodward DB, Botros FT. Dulaglutide versus insulin glargine in patients with type 2 diabetes and moderate-to-severe chronic kidney disease (AWARD-7): a multicentre, open-label, randomised trial. Lancet Diabetes Endocrinol. 2018 Aug;6(8):605-617. doi: 10.1016/S2213-8587(18)30104-9. Epub 2018 Jun 14. PMID 29910024

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a parallel-arm, non-inferiority study. Study treatment continued for up to 52 weeks and participants were randomized in a 1:1:1 ratio to one of the 3 treatment arms: 1.5 milligrams (mg) dulaglutide once-weekly , 0.75 mg dulaglutide once-weekly, or insulin glargine once-daily.
Period: Overall Study
Arm/Group | Insulin Glargine | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide
Started | 194 | 190 | 193
Received at Least One Dose of Study Drug | 194 | 190 | 192
Modified Intent to Treat Population | 186 | 180 | 183
Completed | 163 | 160 | 157
Not Completed | 31 | 30 | 36
Not completed — Adverse Event | 5 | 2 | 8
Not completed — Death | 6 | 7 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Withdrawal by Subject | 14 | 17 | 18
Not completed — Physician Decision | 5 | 2 | 7

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug and had evaluable post-baseline measurements.
Groups:
- Insulin Glargine: Insulin glargine was administered SC at bedtime per a modified forced-titration treat-to-target algorithm. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
- Dulaglutide 0.75 mg: Dulaglutide 0.75 mg administered once weekly as a SC injection. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
- Dulaglutide 1.5 mg: Dulaglutide 1.5 mg administered once weekly as a SC injection. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg | Total
Number analyzed (Participants) | 194 | 190 | 192 | 576
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.41) | 64.7 (8.61) | 64.7 (8.83) | 64.6 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 86 | 88 | 275
  Male | 93 | 104 | 104 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 75 | 78 | 232
  Not Hispanic or Latino | 115 | 115 | 114 | 344
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 17 | 12 | 47
  Asian | 5 | 4 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 26 | 36 | 26 | 88
  White | 137 | 122 | 134 | 393
  More than one race | 6 | 7 | 10 | 23
  Unknown or Not Reported | 1 | 4 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 14 | 9 | 14 | 37
  Hungary | 22 | 19 | 14 | 55
  United States | 61 | 59 | 62 | 182
  Ukraine | 17 | 11 | 12 | 40
  Brazil | 44 | 47 | 50 | 141
  Poland | 1 | 2 | 2 | 5
  Mexico | 19 | 19 | 15 | 53
  South Africa | 14 | 20 | 17 | 51
  Spain | 2 | 4 | 6 | 12
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 88.20 (18.488) | 90.88 (18.301) | 88.14 (16.015) | 89.06 (17.653)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/square meter (kg/m^2)] | 32.39 (5.324) | 33.00 (5.546) | 32.11 (4.841) | 32.50 (5.248)
Hemoglobin A1C (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.56 (0.966) | 8.57 (1.088) | 8.59 (0.860) | 8.57 (0.973)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 18.71 (8.742) | 17.95 (8.788) | 17.57 (8.722) | 18.08 (8.748)
Duration of Chronic Kidney Disease (CKD) Stage 3 or Higher [Mean (Standard Deviation); unit: years] | 3.47 (3.998) | 4.03 (4.854) | 4.18 (5.632) | 3.89 (4.872)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: milliliter/minute/1.73 square meter] | 38.5 (12.99) | 38.3 (12.31) | 38.1 (13.24) | 38.3 (12.83)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least square (LS) means in HbA1c were calculated using a restricted maximum likelihood (REML) based mixed-effects model for repeated measures (MMRM) with the change in HbA1c as the dependent variable and treatment, macroalbuminuria (MA) region, Baseline CKD Severity, week, treatment*week, baseline HbA1c (%), log baseline eGFR (within CKD severity), and participant was the random effect. Covariance structure = Unstructured.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline HbA1c data. Only measurements prior to rescue or study drug discontinuation were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Insulin Glargine: Insulin glargine was administered subcutaneous (SC) at bedtime per a modified forced-titration treat-to-target algorithm. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
- Dulaglutide 0.75 mg: Dulaglutide 0.75 mg was administered once weekly as a SC injection. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
- Dulaglutide 1.5 mg: Dulaglutide 1.5 mg was administered once weekly as a SC injection. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 175 | 149 | 138
percentage of HbA1c | -1.13 (0.12) | -1.12 (0.12) | -1.19 (0.13)
Statistical Analysis 1: Comparison: Insulin Glargine vs Dulaglutide 1.5 mg; Week 26; Test type: Non-Inferiority — Non-Inferiority to Glargine with a 0.4% margin; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.26 to 0.15]
Statistical Analysis 2: Comparison: Insulin Glargine vs Dulaglutide 0.75 mg; Week 26; Test type: Non-Inferiority — Non-Inferiority to Glargine with a 0.4% margin; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.18 to 0.22]

2. Secondary Outcome: Percentage of Participants Whose HbA1c Was <7.0%
Description: Percentage of participants whose HbA1c was <7.0% based on last observation carried forward (LOCF).
Time Frame: 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable post-baseline HbA1c data. Only measurements prior to rescue or study drug discontinuation were used
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 182 | 164 | 152
percentage of participants | 34.6 | 31.7 | 37.5

3. Secondary Outcome: Percentage of Participants Whose HbA1c Was <8.0%
Description: Percentage of Participants whose HbA1c was <8.0% based on last observation carried forward (LOCF).
Time Frame: 26 Weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 182 | 164 | 152
percentage of participants | 75.3 | 72.6 | 78.3

4. Secondary Outcome: Change From Baseline in 8-Point Self-Monitored Plasma Glucose (SMPG)
Description: The daily mean of 8-point SMPG profile at Week 26 is presented. Participants were required to perform two 8-point SMPG profiles over a 1-week period at 5 separate times throughout the study. LS means were calculated using the MMRM model including the corresponding baseline value as a continuous covariate, as well as baseline HbA1c, MA-region, treatment, week, treatment*week, baseline CKD severity, and log baseline eGFR (within CKD severity).The two 8-point SMPG profiles were collected on two non-consecutive days (pre-meal and 2-hour postprandial SMPG x [morning, midday, and evening meals in one day] + bedtime + 5 hours after bedtime).
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline HbA1c and SMPG data. Only measurements prior to rescue or study drug discontinuation were used.
Measure: Least Squares Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 128 | 107 | 102
milligrams/deciliter (mg/dL) | -37.6 (3.41) | -31.7 (3.53) | -33.7 (3.77)

5. Secondary Outcome: Change From Baseline in Fasting Glucose (FG)
Description: LS means were calculated using MMRM with the change in FG as the dependent variable and treatment, MA -region, Baseline CKD Severity, week, treatment*week, baseline FG, baseline HbA1c (%), log baseline eGFR (within CKD severity), and participant was the random effect. Covariance structure = Unstructured
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline HbA1c and FG data. Only measurements prior to rescue or study drug discontinuation were used.
Measure: Least Squares Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 162 | 145 | 132
milligram/deciliter (mg/dL) | -19.1 (6.00) | 17.7 (6.14) | 23.1 (6.50)

6. Secondary Outcome: Change From Baseline in Mean Daily Insulin Lispro Dose
Description: The mean daily insulin was based on a 4-week interval prior to week 26 assessments. LS means were calculated using a REML based mixed-effects model for repeated measures (MMRM) with the change in mean daily insulin as the dependent variable and treatment, MA-region, Baseline HbA1c, baseline mean daily insulin, baseline CKD Severity, week, treatment*week, log baseline eGFR (within CKD severity), and participant was the random effect. Covariance structure = Unstructured.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline HbA1c and insulin lispro dose data. Only measurements prior to rescue or study drug discontinuation were used.
Measure: Least Squares Mean (Standard Error); unit: Units/day (U/day)
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 177 | 154 | 141
Units/day (U/day) | 16.64 (2.76) | 26.16 (2.80) | 18.12 (3.00)

7. Secondary Outcome: Percentage of Participants With Estimated Average Glucose <154 mg/dL
Description: Percentage of Participants With Estimated Average Glucose <154 milligram/deciliter (mg/dL) was based on last observation carried forward (LOCF).
Time Frame: 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable HbA1c and average self-monitored plasma glucose post-baseline data. Only measurements prior to rescue or study drug discontinuation were used.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 134 | 118 | 110
percentage of participants | 64.9 | 52.5 | 56.4

8. Secondary Outcome: Change From Baseline in Serum Creatinine (sCr)
Description: Change from baseline in serum creatinine (sCr) levels after treatment.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received one dose of study drug and had evaluable baseline and post-baseline sCr data.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 176 | 169 | 163
mg/dL | 0.10 [-0.04 to 0.28] | 0.02 [-0.15 to 0.15] | 0.04 [-0.14 to 0.20]

9. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: The change in estimated glomerular filtration rate (eGFR) by using CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline eGFR data.
Measure: Median (Inter-Quartile Range); unit: milliliter/minute/1.73m2 (mL/min/1.73m2)
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 176 | 169 | 163
milliliter/minute/1.73m2 (mL/min/1.73m2) | -2.5 [-6.0 to 1.0] | -1.0 [-4.5 to 3.0] | -1.0 [-5.5 to 3.0]

10. Secondary Outcome: Change From Baseline in Estimated Creatinine Clearance (eCrCl)
Description: Estimated creatinine clearance (eCrCl) was calculated by Cockcroft-Gault [Cockcroft and Gault 1976] equation using baseline estimated lean body weight.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline eCrCl data.
Measure: Median (Inter-Quartile Range); unit: milliliter/minute (ml/min)
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 176 | 169 | 163
milliliter/minute (ml/min) | -2.0 [-4.0 to 0.5] | -1.0 [-3.5 to 2.0] | -0.5 [-4.0 to 2.0]

11. Secondary Outcome: Change From Baseline in Urinary Albumin to Creatinine Ratio (UACR)
Description: The change from baseline in Urinary Albumin to Creatinine Ratio (UACR).
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received one dose of study drug and had evaluable baseline and post-baseline UACR data.
Measure: Median (Inter-Quartile Range); unit: gram/kilogram (g/kg)
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 181 | 175 | 175
gram/kilogram (g/kg) | -1.3 [-71.7 to 62.0] | -11.1 [-147.8 to 33.2] | -10.2 [-180.5 to 53.1]

12. Secondary Outcome: Change From Baseline in Body Weight
Description: LS means were calculated from a REML based MMRM model: Change from Baseline = treatment, week, treatment*Week, MA-region, Baseline HbA1c (%), Baseline Body Weight (kg), Baseline CKD Severity, Log Baseline eGFR (within CKD severity), where participant enters the model as a random effect. Covariance structure = Unstructured.
  •
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline body weight data. Only measurements prior to rescue or study drug discontinuation were used.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 175 | 151 | 140
kilogram (kg) | 1.11 (0.346) | -2.02 (0.357) | -2.81 (0.374)

13. Secondary Outcome: Percentage of Participants With Self-Reported Hypoglycemic Events (HE)
Description: Hypoglycemic events (HE) were classified as severe (defined as an episode requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of ≤3.9 mmol/L (≤70 mg/dL), nocturnal (defined as any hypoglycemic event that occurs between bedtime and waking). The number of self-reported hypoglycemic events was summarized cumulatively at 26 weeks. A summary of other nonserious AEs, and all SAEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through 26 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable post-baseline HE data. Only measurements prior to rescue or study drug discontinuation were used.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 194 | 189 | 190
percentage of participants
  Total Hypo | 71.6 | 50.8 | 43.2
  Documented Symptomatic Hypo | 60.3 | 40.7 | 31.6
  Severe Hypo | 4.1 | 1.1 | 0
  Nocturnal Hypo | 38.1 | 15.9 | 13.2

14. Secondary Outcome: Rate of Hypoglycemic Events
Description: Hypoglycemic events (HE) were classified as total HE rate, documented symptomatic hypoglycemia, severe hypoglycemia, and nocturnal. The 1-year adjusted rate of HEs was summarized cumulatively at 26 weeks. A summary of other nonserious AEs, and all SAEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through 26 Weeks
Population: All randomized participants who had received at least one dose of study drug and had evaluable post-baseline HE rate data. Only measurements prior to rescue or study drug discontinuation were used.
Measure: Mean (Standard Deviation); unit: Events/Participant/Year
Groups:
- Insulin Glargine: Insulin glargine administered SC to be given at bedtime per sliding scale. Participants were instructed to administer their titrated prandial insulin lispro dose SC with the three most significant meals of the day.
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 194 | 189 | 190
Events/Participant/Year
  Total HE Rate | 17.07 (27.70) | 7.76 (20.39) | 5.45 (12.54)
  Documented Symptomatic HE Rate | 11.34 (22.04) | 4.86 (13.37) | 4.19 (11.58)
  Severe HE Rate | 0.10 (0.56) | 0.03 (0.31) | 0.00 (0.00)
  Nocturnal HE Rate | 3.06 (7.26) | 0.73 (2.25) | 0.63 (2.26)

15. Secondary Outcome: Change From Baseline in HbA1c
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. LS means in HbA1c were calculated using a REML based mixed-effects model for repeated measures (MMRM) with the change in HbA1c as the dependent variable and treatment, MA region, Baseline CKD Severity, week, treatment*week, baseline HbA1c (%), log baseline eGFR (within CKD severity), and participant was the random effect. Covariance structure = Unstructured.
Time Frame: Baseline, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 153 | 132 | 130
percentage of HbA1c | -1.00 (0.12) | -1.10 (0.12) | -1.10 (0.13)

16. Secondary Outcome: Percentage of Participants Whose HbA1c is <7.0%
Description: Percentage of participants whose HbA1c was <7.0% based on last observation carried forward (LOCF).
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 182 | 164 | 152
percentage of participants | 29.1 | 33.5 | 32.9

17. Secondary Outcome: Percentage of Participants Whose HbA1c is <8.0%
Description: Percentage of participants whose HbA1c was <8.0% based on last observation carried forward (LOCF).
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 182 | 164 | 152
percentage of participants | 70.3 | 69.5 | 69.1

18. Secondary Outcome: Change From Baseline in 8-Point SMPG
Description: The daily mean of 8-point SMPG profile at Week 52 is presented. Participants were required to perform two 8-point SMPG profiles over a 1-week period at 5 separate times throughout the study. LS means were calculated using the MMRM model including the corresponding baseline value as a continuous covariate, as well as baseline HbA1c, MA-region, treatment, week, treatment*week, baseline CKD severity, and log baseline eGFR (within CKD severity).The two 8-point SMPG profiles were collected on two non-consecutive days (pre-meal and 2-hour postprandial SMPG x [morning, midday, and evening meals in one day] + bedtime + 5 hours after bedtime).
Time Frame: Baseline, 52 Weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 118 | 96 | 102
mg/dL | -40.5 (3.59) | -30.0 (3.75) | -27.2 (3.93)

19. Secondary Outcome: Change From Baseline in FG
Description: as for outcome 5
Time Frame: Baseline, 52 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline HbA1c and FG data. Only measurements prior to rescue or study drug discontinuation were used.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 152 | 132 | 131
mg/dL | -6.4 (6.38) | 20.8 (6.58) | 28.3 (6.87)

20. Secondary Outcome: Change in Mean Daily Insulin Lispro Dose
Description: The mean daily insulin was based on a 4-week interval prior to week 52 assessments. LS means were calculated using a REML based mixed-effects model for repeated measures (MMRM) with the change in mean daily insulin as the dependent variable and treatment, MA-region, Baseline HbA1c, baseline mean daily insulin, baseline CKD Severity, week, treatment*week, log baseline eGFR (within CKD severity), and participant was the random effect. Covariance structure = Unstructured.
Time Frame: Baseline, 52 Weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: U/day
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 159 | 140 | 132
U/day | 16.84 (2.87) | 27.46 (2.93) | 20.05 (3.13)

21. Secondary Outcome: Percentage of Participants With Estimated Average Glucose <154 mg/dL
Description: as for outcome 7
Time Frame: 52 Weeks
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 137 | 122 | 116
percentage of participants | 73.7 | 57.4 | 50.9

22. Secondary Outcome: Change From Baseline in sCr
Description: Change from baseline in sCr levels after treatment.
Time Frame: Baseline, 52 Weeks
Population: All randomized participants who received one dose of study drug and had evaluable baseline and post-baseline sCr data.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 164 | 160 | 157
mg/dL | 0.12 [-0.05 to 0.38] | 0.04 [-0.11 to 0.27] | 0.07 [-0.11 to 0.21]

23. Secondary Outcome: Change From Baseline in eGFR
Description: The change in eGFR by using CKD-EPI equation.
Time Frame: Baseline, 52 Weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m2
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 164 | 160 | 157
mL/min/1.73m2 | -3.3 [-7.5 to 1.0] | -1.5 [-5.5 to 2.5] | -2.0 [-6.0 to 2.5]

24. Secondary Outcome: Change From Baseline in eCrCl
Description: eCrCl was calculated by Cockcroft-Gault [Cockcroft and Gault 1976] equation using baseline estimated lean body weight.
Time Frame: Baseline, 52 Weeks
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 164 | 160 | 157
mL/min | -2.5 [-5.8 to 0.5] | -1.3 [-4.0 to 1.5] | -1.5 [-5.0 to 1.5]

25. Secondary Outcome: Change From Baseline in UACR
Description: The change from baseline in UACR
Time Frame: Baseline, 52 Weeks
Population: All randomized participants who received one dose of study drug and had evaluable baseline and post-baseline UACR data.
Measure: Median (Inter-Quartile Range); unit: g/kg
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 165 | 162 | 159
g/kg | 3.5 [-56.2 to 138.1] | -3.0 [-88.5 to 87.6] | -11.5 [-158.0 to 42.9]

26. Secondary Outcome: Change From Baseline in Body Weight
Description: LS means were calculated from a REML based MMRM model: Change from Baseline = treatment , week, treatment*Week, MA-region, Baseline HbA1c (%), Baseline Body Weight (kg), Baseline CKD Severity, Log Baseline eGFR (within CKD severity), where participant enters the model as a random effect. Covariance structure = Unstructured.
Time Frame: Baseline, 52 Weeks
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 158 | 137 | 132
kg | 1.57 (0.429) | -1.71 (0.448) | -2.66 (0.467)

27. Secondary Outcome: Percentage of Participants With Self-Reported Hypoglycemic Events (HE)
Description: Hypoglycemic events (HE) were classified as severe (defined as an episode requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of ≤3.9 mmol/L (≤70 mg/dL), nocturnal (defined as any hypoglycemic event that occurs between bedtime and waking). The number of self-reported hypoglycemic events was summarized cumulatively at 52 weeks. A summary of other nonserious AEs, and all SAEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through 52 Weeks
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 194 | 189 | 190
percentage of participants
  Total Hypo | 74.7 | 59.8 | 50.0
  Documented Symptomatic Hypo | 63.4 | 48.1 | 40.5
  Severe Hypo | 6.7 | 2.6 | 0
  Nocturnal Hypo | 47.9 | 23.8 | 20.5

28. Secondary Outcome: Rate of Hypoglycemic Events (HE)
Description: HE were classified as total HE rate, documented symptomatic hypoglycemia, severe hypoglycemia, and nocturnal. The 1-year adjusted rate of HEs was summarized cumulatively at 52 weeks. A summary of other nonserious AEs, and all SAEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through 52 Weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Events/Participant/Year
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 194 | 189 | 190
Events/Participant/Year
  Total HE Rate | 14.36 (22.20) | 7.59 (17.81) | 5.82 (13.70)
  Documented Symptomatic HE Rate | 9.62 (17.72) | 4.34 (9.30) | 4.44 (12.23)
  Severe HE Rate | 0.09 (0.37) | 0.03 (0.21) | 0.00 (0.00)
  Nocturnal HE Rate | 2.48 (5.10) | 0.76 (2.09) | 0.70 (2.29)

29. Secondary Outcome: Participants With Events of Allergic/Hypersensitivity Reactions
Description: Participants with Events of Allergic/Hypersensitivity Reactions: Angioedema Standardized MedDRA Query (SMQ), Anaphylactic Reaction SMQ, or Severe Cutaneous Adverse Reactions SMQ
Time Frame: Baseline through 52 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants with events
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 194 | 190 | 192
participants with events
  Angioedema SMQ | 1 | 2 | 2
  Angioedema | 0 | 0 | 1
  Eyelid edema | 0 | 1 | 0
  Face edema | 0 | 1 | 1
  Urticaria | 1 | 0 | 0
  Anaphylactic Reaction SMQ | 1 | 0 | 0
  Circulatory collapse | 1 | 0 | 0
  Severe Cutaneous Adverse Reactions SMQ | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up To Week 52
Description: Safety population included those participants who received at least one dose of study drug.
Arm/Group | Insulin Glargine | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Serious Adverse Events (participants affected / at risk) | 56/194 | 48/190 | 41/192
Other Adverse Events (participants affected / at risk) | 130/194 | 134/190 | 144/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Glargine (N=194) | Dulaglutide 0.75 mg (N=190) | Dulaglutide 1.5 mg (N=192)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 6 (6) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (6)
Chest pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pacemaker generated arrhythmia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (3) | 3 (3) | 3 (3)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 13 (17) | 6 (7) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Iiird nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 5 (5) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 2 (4) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 1/101 (1) | 0/86 (0) | 0/88 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine (N=194) | Dulaglutide 0.75 mg (N=190) | Dulaglutide 1.5 mg (N=192)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 3 (3) | 5 (5)
Constipation (Gastrointestinal disorders) | 6 (6) | 10 (10) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 14 (17) | 30 (37) | 31 (49)
Nausea (Gastrointestinal disorders) | 9 (9) | 27 (38) | 38 (52)
Vomiting (Gastrointestinal disorders) | 9 (9) | 16 (22) | 26 (42)
Oedema peripheral (General disorders) | 15 (16) | 12 (13) | 10 (10)
Influenza (Infections and infestations) | 10 (10) | 15 (18) | 12 (12)
Nasopharyngitis (Infections and infestations) | 12 (15) | 9 (12) | 11 (12)
Sinusitis (Infections and infestations) | 11 (13) | 4 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 20 (26) | 13 (15) | 8 (9)
Urinary tract infection (Infections and infestations) | 19 (25) | 10 (12) | 13 (16)
Blood creatinine increased (Investigations) | 90 (124) | 71 (102) | 74 (106)
Glomerular filtration rate decreased (Investigations) | 26 (29) | 20 (25) | 17 (22)
Weight increased (Investigations) | 16 (18) | 9 (9) | 9 (10)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 5 (6) | 11 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 13 (15) | 8 (10) | 12 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (8) | 10 (10)
Dizziness (Nervous system disorders) | 10 (12) | 11 (12) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 7 (7) | 7 (8)
Hypertension (Vascular disorders) | 20 (20) | 13 (13) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days